CLINICAL TRIAL: NCT07094919
Title: An Cohort Study of Corheart 6 Left Ventricular Assist System for the Treatment of Patients With Advanced Left Heart Failure
Brief Title: Corheart 6: Long-term Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ZX036
Record Dates: First submitted 2025-07-28; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: advanced heart failure; Corheart 6
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corheart 6 Left Ventricular Assist System (Experimental): Subjects with advanced left heart failure despite receiving optimal medical therapy, as per current heart failure management guidelines
  Interventions: Device: Corheart 6 left ventricular assist system

INTERVENTIONS:
Device: Corheart 6 left ventricular assist system — Corheart 6 left ventricular assist system provides circulatory support for patients with advanced left heart failure.

SUMMARY:
This study aims to evaluate the long-term effectiveness and safety of Corheart 6 left ventricular assist system as a treatment for patients with advanced left heart failure. The patients who have received the Corheart 6 treatment since October 2021, or who are planned to received it, will be enrolled until the target sample size meets statistical requirements.

Data collected will include survival status, cardiac function status, quality of life, laboratory parameters and adverse events. The primary endpoint are the composite of survival at 6 months and, separately, at 24 months, defined as survival with device support, bridge to heart transplant and device explantation due to cardiac recovery, without disabling stroke (mRS > 3) or device replacement. Data collection will adhere to the follow-up schedule specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Subject who have undergone Corheart 6 implantation on or after October 1, 2021.
* Body Surface Area (BSA) > 1.0 m2.
* Women of childbearing potential must use agree to use a effective method of contraception for the duration of the study.
* Diagnosis of NYHA Class IV heart failure, refractory to optimal guideline-directed medical therapy (GDMT) (e.g., ACE inhibitors, β-blockers, and diuretics).
* Left Ventricular Ejection Fraction (LVEF) < 30%, with at least one of the following conditions:

  1. Dependence on an intra-aortic balloon pump (IABP), extracorporeal membrane oxygenation (ECMO), or other short-term mechanical circulatory support with an inability to be weaned.
  2. Dependence on continuous intravenous inotropic support.
  3. Meets the diagnostic criteria for cardiogenic shock: blood pressure < 90/60 mmHg, cardiac index < 2.0, pulmonary capillary wedge pressure > 18 mmHg
* Subject or their legally authorized representative agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

* Heart failure caused by unresolved thyroid disease, hypertrophic obstructive cardiomyopathy, pericardial disease, or related conditions.
* Presence of active, uncontrolled infection confirmed through clinical symptoms and laboratory tests.
* Based on the investigator's judgment, presence of technical difficulties that would lead to unacceptable surgical risk.
* Subject is intolerant to anticoagulation or antiplatelet therapy, or cannot receive other perioperative and postoperative treatments deemed necessary by the investigator based on the patient's health condition.
* Require biventricular assist device support.
* Pregnancy.
* Presence of moderate to severe aortic regurgitation or a history of mechanical aortic valve implantation but refuse or is unable to converted to a bioprosthesis or oversewn at the time of LVAD implant.
* History of any organ transplant.
* Presence of unresolved thrombocytopenia or severe coagulopathy, such as disseminated intravascular coagulation (DIC).
* Preoperative total bilirubin (TBIL) > 3.0 mg/dL, serum creatinine (SCr) > 3.0 mg/dL, or requirement for dialysis within 48 hours prior to surgery.
* History of severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, or diagnosed primary pulmonary hypertension.
* Presence of pulmonary embolism within 3 weeks prior to enrollment.
* Pulmonary artery systolic pressure greater than 60 mmHg and meet at least one of the criteria which prove the pulmonary vessels is unresponsive to pharmacologic intervention: a. most recent pulmonary vascular resistance (PVR) ≥ 8 Woods; b. transpulmonary pressure > 20mmHg.
* History of confirmed, untreated abdominal aortic aneurysm (AAA) or thoracic aortic aneurysm (TAA) > 5 cm in diameter.
* Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration.
* Mental illness/disorder, irreversible cognitive dysfunction, or psychosocial issues that may prevent the patient from adhering to the study protocol and the management of the implanted left ventricular assist device, or any condition leading to brain death.
* Presence cancer or other diseases that could limit survival to less than 24 months.
* Participation in any other clinical investigation that is likely to confound study results or affect the study.
* Unforeseen circumstances that the investigator determines to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite survival rate at 6 months. | 6 months
  The composite survival is defined as one of the following criteria, without disabling stroke (modified Rankin Score >3 ), device replacement due to device malfunction, or urgent heart transplant due to device malfunction:
  * heart transplant;
  * explantation for cardiac recovery;
  * survival with device support.
Composite survival rate at 24 months | 24 months

SECONDARY OUTCOMES:
Composite survival rate at 5 years post device implantation | 5 years
NYHA Functional Class | Baseline, 6 months, 24 months, and 5 years post-implantation
6-minute walk test distance | Baseline, 6 months, 24 months, and 5 years post-implantation
EuroQol-5D | Baseline, 6 months, 24 months, 5 years post-implantation
Adverse Events | Up to 5-year post-implantaiton
Reoperation | Up to 5-year post-implantation
Rehospitalization | Up to 5-year post-implantation

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Guangdong
  - the 7Th People'S Hospital of Zhengzhou, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan asia heart hospital, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - the First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Fuwai Hospital, Beijing
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
At this moment the IPD is not yet available for access and will be updated when it is ready.